CLINICAL TRIAL: NCT02956382
Title: Ibrutinib and Venetoclax in Relapsed and Refractory Follicular Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: AbbVie (Industry); Pharmacyclics LLC. (Industry); Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-0014
Record Dates: First submitted 2016-11-02; First posted 2016-11-07 (Estimated); Results first posted 2024-05-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-06

CONDITIONS: Refractory Follicular Lymphoma; Relapsed Follicular Lymphoma
Keywords: Ibrutinib; Venetoclax; Follicular; Refractory; Relapsed; Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Recurrence; Lymphoma | interventions — ibrutinib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase I - Dose Level 0 (Experimental): Ibrutinib (capsule) - 420mg Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Phase I - Dose Level 1 (Experimental): Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Phase I - Dose Level 2 (Experimental): Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 600mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Phase I - Dose Level 3 (Experimental): Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 800mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax
- Phase II Dose (Experimental): The Phase II dose will be the maximum tolerated dose as determined in the Phase I portion.
  Interventions: Drug: Ibrutinib; Drug: Venetoclax

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib is dispensed as a capsule.
  Other Names: PCI-32765
Drug: Venetoclax — Venetoclax is dispensed as a tablet.
  Other Names: ABT-199

SUMMARY:
This is a phase I/II study in which patients will be enrolled in a standard 3+3 design. Once the maximum tolerated dose (MTD) is determined amongst patients with relapsed or refractory grade 1-3a follicular lymphoma, there will be a 17-patient phase II study.

DETAILED DESCRIPTION:
In vitro studies of ibrutinib and venetoclax have noted significant cytotoxicity and synergy in mantle cell lymphoma and chronic lymphocytic leukemia cell lines.Data have demonstrated synergy between the two agents in various other B-cell Non-Hodgkin Lymphoma (NHL) cell lines. The investigators theorize that the combination of ibrutinib and venetoclax will provide dual, yet unique, targeted inhibition for patients with follicular lymphoma, resulting in both significant efficacy and less nonspecific toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory, histologically confirmed follicular lymphoma, grade I, II, or IIIa which requires therapy defined by at least one of the following:

   * Constitutional symptoms
   * Cytopenias
2. High tumor burden (single mass > 7 cm, three masses > 3 cm, symptomatic splenomegaly, organ compression or compromise, ascites, pleural effusion)Must have received at least two prior systemic therapies
3. All risk by FLIPI 0-5 factors (Appendix I)
4. Measurable disease Measurable disease must be present either on physical examination or imaging studies; non-measurable disease alone is not acceptable. Any tumor mass > 1.5 cm is acceptable.

   Lesions that are considered non-measurable include the following:
   * Bone lesions (lesions if present should be noted)
   * Ascites
   * Pleural/pericardial effusion
   * Lymphangitis cutis/pulmonis
   * Bone marrow (involvement by lymphoma should be noted)
5. Adequate hematologic function independent of transfusion and growth factor support for at least 3 weeks prior to screening unless attributable to disease. Defined as:

   * Absolute neutrophil count (ANC) >1000 cells/mm3 (1.0 x 109/L). ANC > 500 cells/mm3 is permissible if due to disease.
   * Platelet count >50,000 cells/mm3 (50 x 109/L) unless attributable to disease. Platelet count > 20,000 cells/mm3 is permissible if due to disease.
   * Hemoglobin >8.0 g/dL.
6. Adequate hepatic and renal function defined as:

   * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN) Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≤ 5 is permissible if due to disease.
   * Bilirubin ≤1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin) Bilirubin ≤3 x ULN is permissible if due to disease.
   * Estimated Creatinine Clearance ≥50 ml/min (Cockcroft-Gault based on actual weight)
7. Prothrombin time (PT)/International normalized ratio (INR) <1.5 x ULN and PTT (aPTT) <1.5 x ULN.
8. Men and women ≥ 18 years of age.
9. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2. (Appendix II)
10. Female subjects who are of non-reproductive potential (i.e., post-menopausal by history - no menses for ≥1 year; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
11. Male and female subjects who agree to use highly effective methods of birth control (e.g., condoms, implants, injectables, combined oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or sterilized partner) during the period of therapy and for 30 days after the last dose of study drug

Exclusion Criteria:

1. Chemotherapy, monoclonal antibody, or small molecule kinase inhibitor less than or equal 21 days prior to first administration of study treatment
2. Prior exposure to a Bruton's tyrosine kinase (BTK) or B-cell lymphoma 2 (BCL-2) inhibitor.
3. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ibrutinib or venetoclax.
4. Known allergy to xanthine oxidase inhibitors and/or rasburicase for subjects at risk for tumor lysis syndrome.
5. History of other malignancies, except:

   * Malignancy treated with curative intent and with no known active disease present for ≥ 3 years before the first dose of study drug and felt to be at low risk for recurrence by treating physician.
   * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   * Adequately treated carcinoma in situ without evidence of disease.
6. Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration [>14 days] of > 20 mg/day of prednisone) within 28 days of the first dose of study drug.
7. Undergone an allogeneic stem cell transplant within the past 1 year.
8. Current or history of graft versus host disease
9. Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
10. Recent infection requiring systemic treatment that was completed ≤14 days before the first dose of study drug.
11. Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.03), grade ≤1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
12. Known bleeding disorders (e.g., von Willebrand's disease) or hemophilia.
13. History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
14. Known HIV infection
15. Active infection with hepatitis C virus (HCV) or hepatitis B virus (HBV).

    • Subjects who are positive for hepatitis B core antibody, hepatitis B surface antigen, hepatitis C antibody, must have a negative polymerase chain reaction (PCR) result for the respective disease before enrollment. Those who are PCR positive will be excluded.
16. Any uncontrolled active systemic infection.
17. Major surgery within 4 weeks of first dose of study drug.
18. Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk.
19. Currently active, clinically significant cardiovascular disease, such as uncontrolled arrhythmia or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification; or a history of myocardial infarction, unstable angina, or acute coronary syndrome within 6 months prior to randomization.
20. Unable to swallow capsules or tablets or malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel, symptomatic inflammatory bowel disease or ulcerative colitis, or partial or complete bowel obstruction.
21. Concomitant use of warfarin or other Vitamin K antagonists.
22. Requires treatment with a strong cytochrome P450 CYP3A4/5 inhibitor. (Appendix V)
23. Richter's transformation confirmed by biopsy.
24. Malabsorption syndrome or other condition precluding enteral route of administration.
25. Known Central nervous system (CNS) involvement by lymphoma
26. Erythema multiforme, toxic epidermal necrolysis, or Stevens-Johnson syndrome
27. Lactating or pregnant.
28. Unwilling or unable to participate in all required study evaluations and procedures.
29. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).
30. Currently active, clinically significant hepatic impairment (greater than or equal moderate hepatic impairment according to the Child Pugh classification (see Appendix IX)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra Ujjani, MD, Study Chair — Seattle Cancer Care Alliance
Locations (3):
- United States (3):
  - Georgetown Lombardi Comprehensive Cancer Center, Washington D.C., District of Columbia
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I - Dose Level 0: Ibrutinib (capsule) - 420mg Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Phase I - Dose Level 1: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Phase I - Dose Level 2: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 600mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Phase I - Dose Level 3: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 800mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Phase II- Dose Level 2: The Phase II dose will be the maximum tolerated dose as determined in the Phase I portion. Phase II Dose = Dose level 2, Ibrutinib (560mg), Venetoclax (600mg).
Period: Overall Study
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase II- Dose Level 2
Started | 3 | 6 | 6 | 1 | 8
Completed | 3 | 6 | 6 | 1 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3 | Phase II Dose | Total
Number analyzed (Participants) | 3 | 6 | 6 | 1 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 5 | 2 | 0 | 5 | 13
  >=65 years | 2 | 1 | 4 | 1 | 3 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 0 | 3 | 7
  Male | 3 | 5 | 3 | 1 | 5 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 2
  Not Hispanic or Latino | 3 | 4 | 5 | 1 | 7 | 20
  Unknown or Not Reported | 0 | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 0 | 1
  White | 1 | 3 | 5 | 1 | 7 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 2 | 0 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D)
Description: The maximum tolerated dose of Ibrutinib and Venetoclax as determined by number of DLTs observed. • If 0/3 DLT is observed, dose escalation will continue to the next upper dose level. • If ≥ 2/3 DLTs are observed, then the dose finding procedure will be terminated.
  • If 1/3 DLT is observed, then 3 additional patients will be enrolled in the same dose level. If no DLT is observed from the additional 3 patients, then dose escalation will continue to the next upper dose level. If any DLT is observed from the 3 additional patients, then the previously lower dose will be chosen as the MTD and the dose finding procedure will be terminated.
Time Frame: Cycle 1 (28 days)
Measure: Number; unit: Dose Limiting toxicities
Groups:
- Phase I - Dose Level 0: Dose Level 0: Ibrutinib (capsule) - 420mg, Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 3 | 6 | 6 | 1
Dose Limiting toxicities | 0 | 1 | 0 | 0

2. Primary Outcome: Dose Level 2 Overall Response Rate
Description: Number of participants on the recommended phase II dose level 2, with a partial or complete response, as determined by the revised Lugano Response Criteria for Non-Hodgkin Lymphoma,
Time Frame: 36 months
Population: Combined Phase I and Phase II participant on RP2D, Dose Level 2
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 2: Recommended Phase II Dose Level = Dose level 2, Ibrutinib (560mg), Venetoclax (600mg).
Arm/Group | Dose Level 2
Number analyzed (Participants) | 14
Participants | 9

3. Secondary Outcome: Pharmacokinetics of Ibrutinib (Cmax) Phase 1
Description: Cmax- Maximiumum concentration of Ibrutinib of subjects in Phase 1.
Time Frame: Cycle 1 (28 days)
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 3 | 3 | 4 | 1
ng/mL
  Cycle 1 Day 1 | 185 (84.8) | 253 (222) | 161 (124) | 227 (227)
  Cycle 1 Day 15 | 155 (4.00) | 195 (109) | 181 (105) | 199 (199)

4. Secondary Outcome: Pharmacokinetics of Ibrutinib (Tmax) Phase 1
Description: Tmax (time to maximum) plasma concentrations of ibrutinib for subjects in phase 1
Time Frame: Cycle 1 (28 days)
Measure: Mean (Full Range); unit: hours
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 3 | 3 | 4 | 1
hours
  Cycle 1 Day 1 | 4 [2 to 4] | 2 [2 to 2] | 2 [1 to 2] | 2 [2 to 2]
  Cycle 1 Day 15 | 2 [2 to 2] | 2 [2 to 2] | 2 [2 to 4] | 2 [2 to 2]

5. Secondary Outcome: Pharmacokinetics of Ibrutinib (AUC) Phase 1
Description: Area Under the Curve (AUC) 0 to 24 hours for subjects in phase 1
Time Frame: Cycle 1 (28 days)
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Phase I - Dose Level 0 | Phase I - Dose Level 1 | Phase I - Dose Level 2 | Phase I - Dose Level 3
Number analyzed (Participants) | 3 | 3 | 4 | 1
ng*h/mL
  Cycle 1 Day 1 | 1340 (570) | 1420 (1020) | 793 (533) | 1980 (1980)
  Cycle 1 Day 15 | 1180 (244) | 1170 (304) | 1250 (912) | 2440 (2440)

6. Secondary Outcome: Number of Participants With Treatment-related Adverse Events as Assessed by CTCAE v4.03
Description: Toxicity (attribute and grade) will be summarized for each dose level (0, 1, 2, 3) for all patients who receive at least one dose of study treatment.
Time Frame: 36 months
Population: All subjects who received dose level 2, regardless of the phase of the trial, phase 1 or phase 2, were combined since the adverse events are by dose level received not phase of the trial.
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 0: Dose Level 0: Ibrutinib (capsule) - 420mg, Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
- Dose Level 1: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 400mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Dose Level 2: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 600mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
- Dose Level 3: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 800mg
  Each medication is taken daily. Treatment cycles are 28 days long.
  Ibrutinib: Ibrutinib is dispensed as a capsule.
  Venetoclax: Venetoclax is dispensed as a tablet.
Arm/Group | Dose Level 0 | Dose Level 1 | Dose Level 2 | Dose Level 3
Number analyzed (Participants) | 3 | 6 | 14 | 1
Participants | 3 | 6 | 14 | 1

ADVERSE EVENTS:
Time Frame: From the time of consent to 30 days after discontinuation of treatment (3.5 years)
Groups:
- Phase 1- Dose Level 0: Ibrutinib (capsule) - 420mg Venetoclax (tablet) - 400mg Each medication is taken daily. Treatment cycles are 28 days long. Ibrutinib: Ibrutinib is dispensed as a capsule. Venetoclax: Venetoclax is dispensed as a tablet.
- Phase 1 - Dose Level 1: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 400mg Each medication is taken daily. Treatment cycles are 28 days long. Ibrutinib: Ibrutinib is dispensed as a capsule. Venetoclax: Venetoclax is dispensed as a tablet.
- Phase 1 - Dose Level 2: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 600mg Each medication is taken daily. Treatment cycles are 28 days long. Ibrutinib: Ibrutinib is dispensed as a capsule. Venetoclax: Venetoclax is dispensed as a tablet.
- Phase 1- Dose Level 3: Ibrutinib (capsule) - 560mg Venetoclax (tablet) - 800mg Each medication is taken daily. Treatment cycles are 28 days long. Ibrutinib: Ibrutinib is dispensed as a capsule. Venetoclax: Venetoclax is dispensed as a tablet.
Arm/Group | Phase 1- Dose Level 0 | Phase 1 - Dose Level 1 | Phase 1 - Dose Level 2 | Phase 1- Dose Level 3 | Phase II- Dose Level 2
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/6 | 2/6 | 0/1 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/3 | 2/6 | 0/6 | 0/1 | 1/8
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 6/6 | 1/1 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1- Dose Level 0 (N=3) | Phase 1 - Dose Level 1 (N=6) | Phase 1 - Dose Level 2 (N=6) | Phase 1- Dose Level 3 (N=1) | Phase II- Dose Level 2 (N=8)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Failure to Thrive, Diarrhea, Nausea, Weight loss
Lung infection (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Pneumonia
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1- Dose Level 0 (N=3) | Phase 1 - Dose Level 1 (N=6) | Phase 1 - Dose Level 2 (N=6) | Phase 1- Dose Level 3 (N=1) | Phase II- Dose Level 2 (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Chest Pressure
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Left ear popping Intermittent
Ear and labyrinth disorders, Other, specify (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Fluid in Left Ear
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — hallowing of eyes
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Vision changes
Retinal vascular disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3) | 5 (5) | 5 (14) | 1 (1) | 6 (12)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Intermittent - Loose stools
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Tar-like stools
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0) — Mouth Sores
Mucositis, oral (Gastrointestinal disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Early Satiety
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) — Lack of appetite
Hemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 5 (8) | 4 (10) | 1 (1) | 3 (8)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (5) | 0 (0) | 2 (3)
Chills (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 3 (4) | 3 (3) | 0 (0) | 3 (4)
Fever (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Flu like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Intermittent night sweats
General disorders and administration site conditions - Other, specify (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Abdominal cramping
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Mild lightheadedness
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Scab discoloration
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Gall Stones
Bronchial infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Influenza A
Investigations - Other, specify (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Elevated PSA
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — COVID-19 Infection
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 2 (3) | 5 (5) | 0 (0) | 2 (2)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Sore in mouth
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (2) | 1 (3) | 1 (2) | 2 (3)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (3) | 1 (2) | 1 (1) | 3 (5)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (1) — Slow wound healing
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 2 (7) | 1 (1) | 3 (5) | 1 (3) | 2 (3)
Platelet count decreased (Investigations) | 2 (3) | 1 (1) | 1 (2) | 1 (1) | 1 (2)
Weight loss (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Muscle Cramps
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — leg cramps
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Shoulder Pain, bilateral
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Wound on finger
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Dupuytren's Contracture
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Discomfort by Tailbone
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cramping in Hands and Feet
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 2 (4) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Nervous system disorders - Other, specify (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Lightheadedness Intermittent
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) — Burning with urination
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Englarged Prostate
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Heavy Menstrual Bleeding
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Rhinitis
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Rhinorrhea, yellow discharge
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 2 (3)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Folliculitis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Skin- nevis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) — Rash
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Blisters on tops of hands
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Cracking of skin
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Tenderness at tip of right toe
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Basal Cell Carcinoma Removal
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/82/NCT02956382/Prot_SAP_000.pdf